CLINICAL TRIAL: NCT02403466
Title: Bundling Effective Resident Handoff Tools to Improve Patient Safety: A Multi-Center Pediatric Residency Quality Improvement Initiative
Brief Title: IIPE-PRIS Accelerating Safe Signouts
Acronym: I-PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Lucile Packard Children's Hospital (Other); University of California, San Francisco (Other); Primary Children's Hospital (Other); St. Louis Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); St. Christopher's Hospital for Children (Other); Walter Reed National Military Medical Center (U.S. Federal Agency); The Hospital for Sick Children (Other); OHSU Doernbecher Children's Hospital (Other)
Responsible Party: Principal Investigator, Christopher Landrigan, Research Director, Children's Hospital Boston Inpatient Pediatrics Service Director, Sleep and Patient Safety Program, Brigham and Women's Hospital Associate Professor of Medicine and Pediatrics, Harvard Medical School, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: X10-08-0392; R18AE000029 (NIH)
Record Dates: First submitted 2011-08-01; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Serious Medical Errors; Resident Sign-out
Keywords: Medical errors; Communication; Resident sign-out
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resident Handoff Bundle (Experimental): bundle of interventions designed to improve handoff, including: training of residents in teamwork and handoff techniques; redesign of verbal handoff processes; implementation of handoff mnemonic (I-PASS); implementation of structured written / computerized handoff tool; faculty training in handoffs
  Interventions: Behavioral: Resident Handoff Bundle

INTERVENTIONS:
Behavioral: Resident Handoff Bundle — 1) team training, 2) verbal mnemonics, and 3) standardization of written/computerized handoff tools

SUMMARY:
Because communication and handoff failures are a root cause of two-thirds of "sentinel events"- serious, often fatal preventable adverse events in hospitals improving handoffs has been identified by AHRQ and the Joint Commission as a priority in nationwide efforts to improve patient safety. Comparative Effectiveness Research on handoff tools and processes has identified specific strategies to improve handoffs and reduce medical errors: 1) team training; 2) verbal mnemonics; and 3) use of written/computerized tools to supplement verbal sign-outs. To accelerate residents' use of CER-based handoff practices and improve patient safety, the investigators are implementing the three inventions above as a Resident Handoff Bundle (RHB) in eight pediatric hospitals in the United States and Canada.

DETAILED DESCRIPTION:
The I-PASS Study was initiated in response to mounting evidence that communication and handoff failures are a root cause of two-thirds of "sentinel events" - serious, often fatal, preventable adverse events in hospitals. The Agency on Healthcare Research and Quality (AHRQ) and Joint Commission have identified improving handoffs in care as a priority in nationwide efforts to improve patient safety. Research on handoff tools and processes has identified team training, introduction of verbal mnemonics, and use of written or computerized tools as strategies to improve handoffs and reduce medical errors. This study was designed to evaluate the effect of a resident handoff bundle (RHB) comprised of these three strategies in addressing medical errors, verbal and written miscommunications, and resident workflow and satisfaction.

The US Department of Health and Human Services granted $3 million in funding, with additional support provided by member institutional and private foundations. A total of nine hospitals in the United States and Canada will serve as data collection sites for the study (see list below). Staggered six-month waves of baseline data collection of medical errors and resident workflow, satisfaction, and miscommunications began in January 2010. Each site has a six-month wash-in period to implement the RHB intervention before embarking upon an additional six months of post-intervention data collection. Analysis and dissemination will begin upon completion of data collection at the last wave of sites in April 2013.

Study Sites:

Children's Hospital Boston (Boston, MA) - Coordinating Site Brigham and Women's Hospital (Boston, MA) - Data Coordinating Center

Lucile Packard Children's Hospital (Palo Alto, CA) UCSF Benioff Children's Hospital (San Francisco, CA) OHSU Doernbecher Children's Hospital (Portland, OR) Primary Children's Medical Center (Salt Lake City, UT) St. Louis Children's Hospital (St. Louis, MO) Cincinnati Children's Hospital Medical Center (Cincinnati, OH) Hospital for Sick Children (Toronto, ON) National Capital Consortium (Washington, DC) St. Christopher's Hospital for Children (Philadelphia, PA)

Study Leadership:

Principal Investigator: Christopher Landrigan, MD, MPH Project Leader: Amy Starmer, MD, MPH

ELIGIBILITY:
Inclusion Criteria:

* The study will also include direct observation of house staff residents on the medical service. While implementation of the RHB itself is a QI protocol, the observation and collection of data from residents is research. We will therefore obtain informed consent from residents for participation in the research related to the effects on their care processes and experiences of implementation of the RHB. Participation will be voluntary.
* All resident physicians rotating through study teams during the two 6 month periods of data collection will be included in the study if informed consent is granted. No resident physicians will be excluded on the basis of age, gender, ethnicity, race, or other demographic features. We anticipate enrolling a maximum of 70 resident physicians per site. This number may be significantly less due to the fact that certain residents may rotate through data collection study units more than once during the study period.

Exclusion Criteria:

* The only exclusion criteria will be residents who do not rotate through study units during the data collection periods

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 875 (Actual)
Dates: Start 2010-09; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Rates of serious medical errors | Continuous collection during data collection phase of study (total of 12 months over an 18 month period matched by time of year (i.e., 6 months pre, 6 months wash-in with no data collection, 6 months post-intervention data collection)

SECONDARY OUTCOMES:
Verbal and written miscommunications | up to 28 months
  Residents will be assessed for 1 month periods at a time, both before and after implementing the intervention. This information will be collected in staggered 18-month intervals across all study sites over the course of a 28 month period.
Time spent by residents gathering and signing out data | up to 28 months
  Residents will be assessed for 1 month periods at a time, both before and after implementing the intervention. This information will be collected in staggered 18-month intervals across all study sites over the course of a 28 month period.
Resident satisfaction with sign-out | up to 28 months
  Residents will be assessed for 1 month periods at a time, both before and after implementing the intervention. This information will be collected in staggered 18-month intervals across all study sites over the course of a 28 month period.
Hospital- and patient-level predictors of implementation success | up to 28 months
  analysis of all outcomes above, cross-referenced with hospital indicator codes and patient severity of illness codes

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Landrigan, MD, MPH, Principal Investigator — Boston Children's Hospital; Amy J Starmer, MD, MPH, Study Director — Oregon Health and Sciences University
Locations (10):
- United States (9):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Primary Children's Medical Center, Salt Lake City, Utah
- Hospital for Sick Children, Toronto, Ontario, Canada